CLINICAL TRIAL: NCT07239362
Title: Culturally Adapted Dialectical Behavior Therapy (DBT) for Mental Health in LMICs: A Randomized Controlled Trial (RCT)
Brief Title: CULTURALLY ADAPTED DIALECTICAL BEHAVIOR THERAPY FOR LOW-MIDDLE-INCOME COUNTRIES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PACTDBT2025
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Borderline Personality Disorder (BPD); Dialectical Behavior Therapy; Emotional Dysregulation; Self Harm; Suicidal and Self-injurious Behavior; Depression Anxiety Disorder
Keywords: BPD; DBT; Self harm; Suicide; Borderline personality; Dialectical behavior therapy; Emotional dysregulation
MeSH Terms: conditions — Borderline Personality Disorder; Self-Injurious Behavior; Suicide

STUDY DESIGN:
Intervention Model Description: This will be a rater-blind RCT to evaluate the feasibility and acceptability of culturally adapted DBT in addition to treatment as usual (TAU) compared with TAU only in Pakistan. This study will employ a pre-post measure and parallel design over 18 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted DBT+Treatment as usual (Experimental): In addition to the usual treatment (TAU), which typically involves pharmacotherapy or supportive counselling from a general physician, participants will receive culturally translated and adapted dialectical behaviour therapy (DBT) materials that fit local cultural and linguistic contexts. Such material will include culturally relevant metaphors, examples, and mindfulness practices. Sessions will be conducted in the form of weekly group skills training (emotion regulation, distress tolerance, interpersonal effectiveness, mindfulness), individual therapy sessions (1 hour/week), and telephone coaching as needed.
  Interventions: Other: Culturally adapted DBT
- Treatment as usual (TAU) only (No Intervention): Participants will only receive standard mental health care available in the region (e.g., medication, supportive counselling), usually from a general physician. TAU in Pakistan largely consists of pharmacological treatment with medication and follow-up in an outpatient basis.

INTERVENTIONS:
Other: Culturally adapted DBT — Participants will receive culturally translated and adapted dialectical behaviour therapy (DBT) materials that fit local cultural and linguistic contexts. Such material will include culturally relevant metaphors, examples, and mindfulness practices. Sessions will be conducted in the form of weekly group skills training (emotion regulation, distress tolerance, interpersonal effectiveness, mindfulness), individual therapy sessions (1 hour/week), and telephone coaching as needed.
  Arms: Culturally adapted DBT+Treatment as usual

SUMMARY:
The study aims to assess the efficacy of culturally adapted dialectical behaviour therapy (DBT) for addressing emotional dysregulation in a low- and middle-income country, as well as to evaluate the impact of DBT on secondary outcomes such as borderline personality traits, self-harm or suicide, depression, anxiety, and individuals' functioning and disability.

Through a rigorous Randomised Controlled Trial (RCT), the research seeks to assess how cultural adaptations of dialectical behaviour therapy improve its applicability, engagement, and outcomes in diverse socio-cultural settings, contributing to more accessible and effective mental health interventions in resource-limited regions.

DETAILED DESCRIPTION:
DBT has proven successful in high-income countries; its application in low- and middle-income countries (LMICs) is limited despite the significant mental health burden in these regions. Mental health challenges in LMICs are further compounded by socio-cultural, economic, and infrastructural barriers, highlighting the need for culturally sensitive adaptations of evidence-based therapies. Culturally adapted DBT involves modifying therapeutic components to align with local norms, values, and language, while maintaining its core strategies, including mindfulness, emotion regulation, interpersonal effectiveness, and distress tolerance. Randomised Controlled Trials (RCTs) are essential to evaluate the feasibility, acceptability, and efficacy of such culturally tailored interventions, helping bridge the mental health treatment gap in LMICs. The current study aimed to evaluate the feasibility, acceptability, and clinical effectiveness of a culturally adapted Dialectical Behaviour Therapy (DBT) intervention for addressing mental health challenges in low- and middle-income countries (LMICs) as compared to treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-45 years
* Adults who are diagnosed with or have significant traits of borderline personality disorder (BPD)
* Adults who are willing to provide written informed consent

Exclusion Criteria:

* Severe psychiatric comorbidity (e.g., active psychosis, substance use, etc.)
* Acute medical conditions interfering with participation
* Lack of basic reading and writing, or any learning disability

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Emotional dysregulation | 18 Months
  As measured through participants' scores on the Difficulties in Emotion Regulation Scale-16 item version (DERS-16)
Self-harm or suicide | 18 months
  As measured through the participants' scores on the Self-Harm Inventory, as well as the presence of any suicide attempt in participants' history

SECONDARY OUTCOMES:
Borderline traits | 18 months
  As assessed through participants' scores on the Gul Mahmood Borderline Personality Traits Scale (GMBPTS)
Depression and anxiety | 18 months
  As measured through participants' scores on Hospital Anxiety and Depression Scale (HADS)
Functioning and disability | 18 months
  As assessed through the WHO Disability Assessment Schedule (WHODAS 2.0)

CONTACTS AND LOCATIONS:
Overall Officials: Mirrat G. Butt, PhD, Principal Investigator — PACT
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No